CLINICAL TRIAL: NCT06131034
Title: Does Perioperative Music Prevent Sleep Disturbances in Hospitalized Surgical Patients
Acronym: DREAMERS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, C. Verhoef, Prof. Dr. C. Verhoef, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL78543.078.21
Record Dates: First submitted 2023-09-06; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Sleep
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental)
  Interventions: Other: Music
- Control group (No Intervention)

INTERVENTIONS:
Other: Music — Participant in the intervention group will receive music interventions perioperatively.
  Arms: Music group

SUMMARY:
Sleep disturbances are known to be a prevalent problem in hospitalized, surgical patients, which is of importance since sleep disturbances can lead to a range of negative health outcomes. Music interventions have shown potential in improving sleep quality. Unfortunately, the studies on the effect of music on sleep in surgical patient populations are still scarce and of low quality. Therefore, the aim of this study is to study the effect of music on sleep quality in oncological, gastro-intestinal surgical patients in the form of a randomized controlled trial. Participants will be divided in 2 groups, a music group and a control group, where the music group will receive music interventions perioperatively. The researchers will compare both groups to see if there is a difference in sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients undergoing major elective abdominal surgery for malignant disease, including, but not limited to: Esophageal, gastric, colorectal, hepatic, pancreatic, gynecological and urological surgical procedures.
* Sufficient knowledge of the Dutch language.
* Communicable and able to assess the questionnaires
* Written informed consent acquired from the patient.

Exclusion Criteria:

* Patients with severe hearing impairment (defined as no or barely verbal communication possible).
* The patient is expected to be transferred to another hospital postoperatively.
* Participation in another study that may possibly intervene with the outcome measures. (e.g. in trial use of sleep medication, interventions regarding sleep quality or quantity or similar procedures)
* Assessment of primary outcome is not possible.
* Inability or unwillingness to receive the music intervention.
* Inability to wear the actigraphy device, or inability to perform actigraphy measurement due to paralysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality assessed using a questionnaire | On the morning of day 2, 3 and 4 at the surgical ward
  Using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep disturbance questionnaire, raw summary score

SECONDARY OUTCOMES:
Subjective sleep quantity | During the (possible) intervention period, until day 5 postoperatively
  Using the adapted Consensus Sleeping Diary
Objective sleep assessment | During the (possible) intervention period, until day 5 postoperatively
  Measured with an actigraphy device
Music listening during study period | During the (possible) intervention period, until day 5 postoperatively
  Using a diary
Anxiety | Every morning during the (possible) intervention period, until day 5 postoperatively
  Using the The State-Trait Anxiety Inventory-6 (STAI-6), 20-80, with a high score being a worse outcome
Subclinical stess using | At baseline and at the end of the (possible) intervention period, at day 5 postoperatively
  Using the Subclinical Stress Symptoms Questionnaire (SSQ-25).
Postoperative quality of recovery using a questionnaire | At baseline, at the end of the (possible) intervention period (from start of study until day 5 postoperatively) and 30 days after discharge
  Quality of Recovery-40 score (QOR-40)
Patient satisfaction using a self-made questionnaire | At the end of the study period, 30 days after discharge
  A Likert scale will be used, 0 -10, with a higher score meaning a more satisfied feeling regarding the hospital admittance.
Music preference and importance in daily life | At baseline
  Using a questionnaire with use of multiple chose questions and a Likert scale, 0 - 10, with a higher score resulting in a more positive attitude towards music
Cost consequences and cost-effectiveness | 30 days after discharge
  Using the Institute for Medical Technology Assessment (iMTA) medical consumption questionnaire and the iMTA productivity loss questionnaire
Cost consequences and cost-effectiveness | 30 days after discharge
  Using the Institute for Medical Technology Assessment (iMTA) productivity loss questionnaire
Quality of life score | At baseline, at the end of the (possible) intervention period (from start of study until day 5 postoperatively) and 30 days after discharge
  Using the EuroQol-5dimension-5length (EQ-5D-5L), with a score of 0 - 100, where a higher score
Delirium incidence | During the entire hospital stay surrounding the surgery, up to day 30 postoperatively.
  Delirium Observation Scale per day and delirium diagnosis (defined as diagnosis by clinician)

OTHER OUTCOMES:
Area of residence | At baseline
  Using postal code of current address
General medication use (incidence and concentration) | Before and during admittance, retrospectively, with a maximum of day 30 postoperatively
  Medication use that could be of influence on sleep quality
Physical parameter, bloodpressure | During the entire hospital stay surrounding the surgery, up to day 30 postoperatively.
  in mm/Hg
Physical parameter, pulse rate | During the entire hospital stay surrounding the surgery, up to day 30 postoperatively.
  beats/min
Physical parameter, respiratory rate | During the entire hospital stay surrounding the surgery, up to day 30 postoperatively.
  Resp/min
Perioperative complications | During the entire hospital stay surrounding the surgery, up to day 30 postoperatively.
  Number of patients with medical complications, and grading of these complications using Clavien Dindo and the Comprehensive Complication Index (CCI)
Clinical information checklist | During the entire hospital stay surrounding the surgery, up to day 30 postoperatively.
  Information about type of surgery, selected medical history, age, gender, hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: C. Verhoef, Professor, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stoop JM, Geensen R, Louter M, Poley MJ, Verhoef C, Jeekel J, Klimek M. The DREAMERS-trial: A randomized controlled trial protocol addressing the use of perioperative music to prevent sleep disturbances in hospitalized surgical patients. Contemp Clin Trials. 2025 Dec;159:108129. doi: 10.1016/j.cct.2025.108129. Epub 2025 Oct 24. PMID 41326266